CLINICAL TRIAL: NCT00243191
Title: Study of a Short Course of Neoadjuvant Gleevec (Imatinib Mesylate) in Dermatofibrosarcoma Protuberans
Brief Title: Neoadjuvant Imatinib in Dermatofibrosarcoma Protuberans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SARC004; NCT00176709 (obsolete NCT alias)
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-02

CONDITIONS: Dermatofibrosarcoma Protuberans
Keywords: newly diagnosed or recurrent
MeSH Terms: conditions — Dermatofibrosarcoma; Recurrence | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- imatinib mesylate (Other)
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate — 400 mg orally twice a day for 10 - 14 days
  Other Names: Gleevec

SUMMARY:
The purpose of this study is to examine the effect of imatinib on dermatofibrosarcoma protuberan tumors.

ELIGIBILITY:
Inclusion criteria:

1. Patients ≥ or equal to 18 years of age.
2. Suspected or documented diagnosis of dermatofibrosarcoma protuberans (DFSP). Patients with suspected diagnosis of DSFP must have DFSP confirmed by pathology at the local institution prior to dispensing and the start of imatinib.
3. Patient is medically able to undergo surgical resection of the DFSP and resection of the DFSP is recommended for clinical management of the disease.
4. Patient has at least one site of measurable (macroscopic) disease.
5. Performance status 0, 1 or 2 Eastern Cooperative Oncology Group (ECOG) (see Section 7.1).
6. Adequate end organ function, defined as the following:

   total bilirubin < 1.5 x institutional upper limit of normal (ULN), SGOT and SGPT < 2.5 x UNL, creatinine < 1.5 x ULN, absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L.
7. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
8. Written, voluntary informed consent.

Exclusion criteria:

1. Patients who will receive radiation therapy to the site of DFSP prior to resection.
2. Patients with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria (i.e., congestive heart failure, myocardial infarction within 6 months of study).
3. Female patients who are pregnant or breast-feeding.
4. Patients who have a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection) that may worsen because of imatinib.
5. Patients who have known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
6. Patients who have a known diagnosis of human immunodeficiency virus (HIV) infection.
7. Patients who have received chemotherapy within 4 weeks prior to study entry.
8. Patients who have had a major surgery within 2 weeks prior to study entry. Incisional biopsy or partial excision of dermatofibrosarcoma protuberans to establish the diagnosis and/or to collect pretreatment tumor tissue does not qualify as major surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Schuetze, MD, PhD, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Pennsylvania Onc/Hem Assoc., Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: SARC Website — http://www.sarctrials.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period began May 1, 2006 and was completed July 22, 2009. There were 5 SARC sites participating. SARC sites are primarily academic institutions with Sarcoma programs.
Period: Overall Study
Arm/Group | Imatinib
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: To Collect Matched Tumor Tissue of Trial Participants With Dermatofibrosarcoma Protuberans Before and After Treatment With Imatinib for Future Use in cDNA Microarray and Tissue Array Studies.
Description: To obtain matched tumor tissue samples of trial participants dermatofibrosarcoma protuberans (DFSP)for the purpose of determining whether imatinib mesylate affects autocrine/paracrine stimulated signal transduction through the platelet-derived growth factor receptor pathway in DFSP by comparing the level of phosphorylated platelet-derived growth factor receptor beta (PDGFRB) in DFSP after up to 2 weeks of treatment with imatinib to the level of phosphorylated PDGFRB pre-treatment.
Time Frame: Prior to and after 2-weeks of imatinib therapy
Population: Population of paired tissue samples collected from patients with confirmed diagnosis of dermatofibrosarcoma protuberans. Tissue sample will be considered evaluable if there is adequate pre-treatment and on-treatment tumor tissue available for the proposed molecular studies, and resection of DFSP was completed after receiving imatinib.
Measure: Number; unit: paired tumor tissue samples
Arm/Group | Imatinib
Number analyzed (Participants) | 18
paired tumor tissue samples | 18

ADVERSE EVENTS:
Time Frame: 3 years, 6 months
Arm/Group | Imatinib
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib (N=18)
chest pain (Cardiac disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
infection (Skin and subcutaneous tissue disorders) | 1 (1)
pain (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Dermatofibrosarcoma protuberans (DFSP)is a rare tumor type. During the the trial the drug manufacturer obtained approval for DSFP indication.The other limitation is limited funding; SARC is actively seeking funding for secondary outcome goal 12/2012.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less